CLINICAL TRIAL: NCT06773962
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of TB006 in Participants With Parkinson's Disease
Brief Title: A Phase 2a Multicenter Clinical Trial of TB006 in Participants With Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TrueBinding, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TB006PD2101
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease (PD)
Keywords: PD; TB006; Monoclonal Antibody; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — TB006

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TB006 (Experimental): Participants will receive TB006 via intravenous (IV) infusion.
  Interventions: Drug: TB006
- Placebo (Placebo Comparator): Participants will receive placebo via IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TB006 — IV infusion.
  Arms: TB006
Drug: Placebo — IV infusion.
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to assess the efficacy of TB006 in improving motor function and to assess the safety of TB006 in participants with Parkinson's Disease (PD).

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily agree to participate in this study and sign an Institutional Review Board (IRB)-approved informed consent form (ICF) prior to performing any of the screening procedures.

   Parkinson's Disease Related Criteria:
2. Diagnosis of Parkinson's disease (PD) with motor symptom improvement from levodopa, if applicable.
3. Less than 5 years from the initial PD diagnosis, at the time of ICF.
4. Early-stage PD, with mild symptoms based on standard clinical staging in OFF state.
5. Participants who are on immediate-release levodopa-carbidopa/benserazide.

   Other Health Related Criteria
6. No active cancer, unless in remission for ≥10 years without ongoing treatment, except fully removed basal cell carcinoma.
7. Free of significant health issues that might interfere with study participation.

   Other Criteria/Social Circumstances
8. Negative screening for illegal drugs (excluding cannabis), with willingness to abstain during the study and avoid cannabis or alcohol effects during visits.

Exclusion Criteria:

Parkinsons's Disease Related Criteria

1. History of sudden, unexpected PD medication OFF episodes.
2. Severe motor complications or disabling symptoms that may impact study involvement.

   Other Health Related Criteria
3. Any condition or health concern deemed a safety risk or likely to interfere with study results.
4. Severe psychiatric disorders, including psychosis or substance addiction.
5. Allergies or sensitivities to specific study-related treatments or substances.
6. Any prior history of a severe infusion reaction.

   Other Criteria/Social Circumstances
7. Pregnancy, breastfeeding, or plans for pregnancy or ova donation during or shortly after the study.
8. Recent use of investigational drugs or therapeutic antibodies.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Parkinson's Disease Rating Scale Score | Baseline to 28 weeks
Number of Participants Experiencing Adverse Events | 28 weeks
Number of Participants Experiencing Serious Adverse Events | 28 weeks

SECONDARY OUTCOMES:
Change from Baseline in Parkinson's Disease Rating Scale Sub-score | Baseline to 28 weeks
Change from Baseline in Patient Perceived Severity of Disease | Baseline to 28 weeks
Change from Baseline in Clinician Perceived Severity of Disease | Baseline to 28 weeks

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Parkinson's Research Centers of America - Orange County, Aliso Viejo, California
  - Parkinson's Research Centers of America - Palo Alto, Palo Alto, California
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - University of South Florida Parkinson's and Movement Disorders Center, Tampa, Florida
  - Consultants in Neurology, Ltd, Northbrook, Illinois
  - Josephson Wallack Munshower Neurology - Southeast, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Quest Research Institute, Farmington Hills, Michigan
  - Parkinson's Research Centers of America - Long Island, Commack, New York
  - NYU Langone Health, Patchogue, New York
  - Oregon Health & Science University, Portland, Oregon
  - Central Texas Neurology Consultants, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No